CLINICAL TRIAL: NCT00870662
Title: A Feasibility Study of the Automated Fluid Shunt (AFS) for Automated Ascites Removal
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NovaShunt AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2008-AAR-001
Record Dates: First submitted 2009-03-25; First posted 2009-03-27 (Estimated); Last update posted 2011-12-19 (Estimated); Status verified 2011-12

CONDITIONS: Refractory Ascites
MeSH Terms: conditions — Ascites

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Automatic Fluid Shunt (Experimental)
  Interventions: Device: AFS System

INTERVENTIONS:
Device: AFS System — AFS System with patient specific flow rate

SUMMARY:
The purpose of this study is to determine whether the Automatic Fluid Shunt (AFS) can reduce the number of paracentesis procedures in patients with refractory ascites.

ELIGIBILITY:
Inclusion Criteria:

* Female or male patients ≥ 18 years of age
* Removal of at least 10 L of ascites in the preceding 2 months for symptom relief
* Failure to respond to a maximum of 160 mg/d of furosemide and 400 mg/d of spironolactone (or equivalent doses of loop-acting and distal-acting diuretics), or intolerance to high dose diuretics because of hyponatremia, hyperkalemia, or other side-effects
* Dietary sodium restriction <90 mcg/d.
* Serum creatinine levels of less than 1.8 mg/dL for at least 7 days before study entry.
* Total bilirubin levels of less than 3 mg/dL.
* Expected survival of greater than 6 months
* Written informed consent

Exclusion Criteria:

* Presence of recurring systemic or local infection, such as peritonitis, urinary tract infection, or abdominal skin infection.
* Presence of peritoneal carcinomatosis
* Evidence of extensive ascites loculation
* Obstructive uropathy
* Coagulopathy that could not be corrected to a prothrombin time INR <1.8,
* Thrombocytopenia that could not be corrected to a platelet count greater than 60,000/mm3
* Any other clinically significant disease that could be adversely affected by study participation judged by the Investigator
* Any condition requiring emergency treatment
* Pregnancy
* Inability to obtain informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2008-12; Primary Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Number of paracentesis procedures required | 6 month

CONTACTS AND LOCATIONS:
Locations (2):
- Czechia (2):
  - Vseobecna fakultni nemocnice v Praze, Prague, Prague
  - IKEM, Prague